CLINICAL TRIAL: NCT04604457
Title: Impact of Predictive Modeling on Time to Palliative Care in an Outpatient Primary Care Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rachel D. Havyer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 20-005977
Record Dates: First submitted 2020-10-14; First posted 2020-10-27 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Palliative Care
Keywords: machine learning; predictive model; palliative care

STUDY DESIGN:
Intervention Model Description: Step-wedge design with 7 wedges: the first wedge has all primary care teams in the standard of care arm; every six weeks one or two care teams switch to the intervention arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Palliative care specialists would not reach out to primary care providers. Palliative care needs would be met via existing mechanisms.
- Predictive Model (Experimental): Palliative care specialists review recommendations from the predictive model and contact a patient's primary care provider (PCP) when appropriate to recommend a palliative care consult.
  Interventions: Other: Palliative care contacts primary care

INTERVENTIONS:
Other: Palliative care contacts primary care — Palliative care specialist reaches out to primary care to recommend a palliative care consult. If the primary care provider agrees, he/she will write an order for a palliative care consult.
  Arms: Predictive Model

SUMMARY:
A machine learning algorithm will be used to accurately identify patients in certain primary care units who may benefit from palliative care consults.

DETAILED DESCRIPTION:
A machine learning algorithm will be used to accurately identify patients in certain primary care units who may benefit from palliative care consults. These patients will be presented weekly to a palliative care specialist in a custom user interface. The palliative care specialist will reach out to primary care teams if she determines that the patient would benefit from palliative care. If the primary care provider agrees, he/she would write a palliative care consult order for the patient. The goal is to reduce the time to palliative care for these patients, who may not have been identified as quickly without the algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient assigned to a primary care unit from July 2020 to June 2021.
* Weekly the palliative care specialists will select patients by looking at patients in sorted order starting with the highest score and proceeding down the list and evaluating each patient for exclusion criteria.

Exclusion Criteria:

* Patients that have been seen by Palliative care will be excluded for 75 days
* Patients under the age of 18 years.
* Patients currently enrolled with hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127070 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Timely identification for need of palliative care | Through study completion, an average of 1 year
  Time to electronic record of consult by the palliative care team in the outpatient setting

SECONDARY OUTCOMES:
Number of palliative care consults | Through study completion, an average of 1 year
  Number of palliative care consults that occurred on intervention and standard of care arms
Number of advanced care planning notes documented in the EHR | Through study completion, an average of 1 year
  Number of advanced care planning notes documented in the EHR on both arms
Number of billing codes for palliative care | Through study completion, an average of 1 year
  Number of ICD-10 billing codes for palliative care on both arms
Positive predictive value of screened patients | Through study completion, an average of 1 year
  Percentage of screened patients that received palliative care consults
Percent of patients who are eligible for ECH based palliative care | Through study completion, an average of 1 year
  Percent of patients who are eligible for employee/community health (ECH) based palliative care compared to the Palliative Care Clinic.
Percent agreement between Palliative Care and Primary Care and average time between Primary Care Contact and Response | Through study completion, an average of 1 year
  Agreement statistics (percent agreement and Kappa statistics) between Palliative Care and Primary Care and descriptive statistics (mean, etc.) on time between primary care contact and response.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Havyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinzen EP, Wilson PM, Storlie CB, Demuth GO, Asai SW, Schaeferle GM, Bartley MM, Havyer RD. Impact of a machine learning algorithm on time to palliative care in a primary care population: protocol for a stepped-wedge pragmatic randomized trial. BMC Palliat Care. 2023 Feb 3;22(1):9. doi: 10.1186/s12904-022-01113-0. PMID 36737744
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials